CLINICAL TRIAL: NCT00777777
Title: The eSVS(TM)Mesh External Saphenous Vein Support Trial
Brief Title: The eSVS (TM) Mesh External Saphenous Vein Support Trial
Acronym: eSVS
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Kips Bay Medical, Inc. (Industry); Transmedic Pte Ltd, Singapore (Unknown)
Responsible Party: Uwe Klima, MD, PhD, National University Hospital Singapore
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DSRB-C/08/149
Record Dates: First submitted 2008-10-20; First posted 2008-10-22 (Estimated); Last update posted 2008-10-22 (Estimated); Status verified 2008-10

CONDITIONS: Coronary Artery Disease
Keywords: multi-vessel, therapy, surgery, CABG
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Either the Circumflex Coronary Artery or the Right Coronary Artery will receive the mesh supported vein graft and the native saphenous vein as second and control graft.
  Interventions: Device: eSVS, saphenous vein supporting mesh

INTERVENTIONS:
Device: eSVS, saphenous vein supporting mesh — Surgical coronary artery bypass grafting to the right coronary artery and the circumflex coronary artery with saphenous vein grafts, one will be supported by the eSVS(TM).
  Other Names: eSVS™; Kips Bay Medical

SUMMARY:
Prospective, multi-center, randomized, controlled (patients as their own control) trial on an external mesh device (eSVS™, Kips Bay Medical) supporting saphenous vein grafts for coronary bypass graft surgery in patients with multi-vessel coronary heart disease.

DETAILED DESCRIPTION:
The objective of the eSVS™ Mesh Saphenous Vein Support Trial is to prospectively evaluate the clinical safety and efficacy of the eSVS™ Mesh for the treatment of Saphenous Vein Graft (SVG) Coronary artery bypass grafting (CABG) versus SVG CABG without an eSVS™ Mesh.

The eSVS™ Mesh External Saphenous Vein Support Trial is a prospective, multi-center, randomized, controlled trial enrolling up to 120 patients with multi-vessel coronary artery disease who require SVG CABG of the Right Coronary Artery and the Circumflex Artery due to atherosclerotic coronary artery disease. Patients will serve as their own control (patients will be randomized to either:

1. SVG+eSVS™ Mesh at Right Coronary Artery and SVG at Circumflex Artery or
2. SVG at Right Coronary Artery and SVG+eSVS™ Mesh at Circumflex Artery).

Clinical follow-up assessments consisting of a physical exam, laboratory testing, medication review, and adverse event monitoring for all enrolled patients will be performed at 30 days, 6 months and 12 months. In addition, the 12 month follow-up assessment will include angiography.

The investigational device being evaluated in this clinical trial is an External Saphenous Vein Support device, the eSVS™ Mesh.

The eSVS™ Mesh is an extravascular prosthesis consisting of a highly flexible, semi-compliant knitted nitinol mesh tube that is placed over the patient's saphenous vein graft (SVG) during coronary artery bypass grafting (CABG). The eSVS™ Mesh is designed to:

* provide radial support to the vein to prevent graft dilatation
* reduce the vein graft diameter to more closely match target coronary artery diameter
* provide a more uniform lumen
* improve blood flow characteristics
* mitigate the development of intimal hyperplasia and graft stenosis

The eSVS™ Mesh has compliance characteristics comparable to native internal thoracic arteries. Since the eSVS™ Mesh vascular prosthesis is made of nitinol, it is highly kink resistant.

ELIGIBILITY:
Inclusion Criteria:

1. require on-pump SVG CABG of the Right Coronary Artery and the Circumflex Artery due to atherosclerotic coronary artery disease, with ≥ 75% stenosis in each of these vessels
2. have appropriately sized and accessible target coronary arteries, with a minimum diameter of 1.5 mm and a lack of calcification at the anastomotic site
3. are able to give their informed written consent
4. are ≥ 21 years of age

Exclusion Criteria:

1. no appropriate target coronary vessel
2. discreet attachment of each SVG to the aorta is not possible (non-consecutive or "jump" grafts are excluded)
3. concomitant non-CABG cardiac procedure
4. prior peripheral vascular or cardiac surgery
5. prior stroke
6. history of atrial fibrillation
7. diffuse peripheral vascular disease
8. age > 80
9. LVEF < 30% at time of enrollment
10. Insulin-dependent diabetes
11. concurrent participation in another trial
12. concomitant life-threatening disease likely to limit life expectancy to less than 2 years
13. contra-indications to on-pump CABG with cardioplegic arrest (calcified aorta, calcified coronaries, small target vessels)
14. emergency CABG surgery
15. inability to tolerate or comply with normal post-surgical drug regimen (antiplatelet plus statin)
16. taking warfarin or clopidogrel at the time of surgery
17. inability to comply with required follow-ups, including angiography imaging methods
18. patient is pregnant or intends on becoming pregnant in the next 12 months

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-06 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Primary Efficacy Endpoint: The primary endpoint of the trial is percent stenosis of Study Vessels, assessed by angiography at 12 months following surgery | 12 months
Primary Safety Endpoint: The occurrence of the composite of total mortality, stroke, MI (Q wave and non-Q wave), or coronary revascularization (i.e. coronary artery bypass surgery or percutaneous coronary intervention) at 30 days post surgery | 12 months

SECONDARY OUTCOMES:
The occurrence of the composite of total mortality, stroke, MI (Q wave and non-Q wave), or coronary revascularization (i.e. coronary artery bypass surgery or percutaneous coronary intervention) at discharge, 6 months and 12 months post surgery | 12 months
Per-patient incidence of vein graft failure/occlusion | 12 months
Per-graft incidence of vein graft failure/occlusion | 12 months
Rates of graft failure due to characterization of anastomotic site failure vs. graft failure | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Uwe Klima, MD, PhD, Principal Investigator — Department of Cardiac, Thoracic and Vascular Surgery, National University Hospital Singapore
Locations (1):
- Department of Cardiac, Thoracic and Vascular Surgery, National University Hospital Singapore, Singapore, Singapore

REFERENCES:
- [Background] Mehta D, George SJ, Jeremy JY, Izzat MB, Southgate KM, Bryan AJ, Newby AC, Angelini GD. External stenting reduces long-term medial and neointimal thickening and platelet derived growth factor expression in a pig model of arteriovenous bypass grafting. Nat Med. 1998 Feb;4(2):235-9. doi: 10.1038/nm0298-235. PMID 9461200
- [Background] Klesius AA, Konerding MA, Knez P, Dzemali O, Schmitz-Rixen T, Ackermann H, Moritz A, Kleine P. External stenting with a new polyester mesh reduces neointimal hyperplasia of vein grafts in a sheep model. Int J Artif Organs. 2007 Oct;30(10):930-8. doi: 10.1177/039139880703001011. PMID 17992655